CLINICAL TRIAL: NCT02857179
Title: Prospective Cohort Study Monitoring Patients Undergoing Bariatric Surgery
Brief Title: Study of Bariatric Surgery
Acronym: BARIASURG
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0504
Record Dates: First submitted 2016-07-27; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Bariatric Surgery
Keywords: bariatric surgery; follow-up; weight loss; complications; comorbidities evolution
MeSH Terms: conditions — Weight Loss | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: bariatric surgery — gastric bypass Or gastric banding Or Biliopancreatic diversion with duodenal switch Or sleeve gastrectomy Or endoscopic procedure (Endobarrier,…)

SUMMARY:
The aim of this cohort study is to collect prospectively clinical data on all the patients admitted in the investigators department for bariatric surgery or for any complication of a bariatric procedure. The investigators goal is not only to improve the follow-up but also to assess and publish the investigators results regarding weight loss and the complication rate.

ELIGIBILITY:
Inclusion Criteria:

* History of bariatric surgery procedure

Exclusion Criteria:

* Patients < 16 years
* Patients > 80 years

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Obese patients (BMI > 30) or patients admitted for a bariatric surgery complication
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2007-11; Primary Completion 2032-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Weight loss in kg | Before surgery (Day 0) and After surgery (every year, up to 25 years or loss to follow-up)
Weight loss in kg/m² | Before surgery (Day 0) and After surgery (every year, up to 25 years or loss to follow-up)
Excess Weight Loss | Before surgery (Day 0) and After surgery (every year, up to 25 years or loss to follow-up)
% weight loss | Before surgery (Day 0) and After surgery (every year, up to 25 years or loss to follow-up)

SECONDARY OUTCOMES:
type of surgical procedure | at the time of surgery (Day 1)
  gastric bypass, sleeve gastrectomy, gastric banding, biliopancreatic diversion, redo surgery, endoscopic procedure…
age | before surgery (Day 0)
  demographic data: age
gender | before surgery (Day 0)
  demographic data: gender
Type of comorbidities | before surgery (Day 0)
  demographic data: comorbidities (diabetes, arterial hypertension, sleep apnea, dyslipidemia)
surgical complications | per and postoperative (up to 25 years or loss to follow-up)
  leaks, hemorrhage, phlebitis, pulmonary embolism, nutritional deficiencies, occlusions,…
dose of insulin | after surgery (up to 25 years or loss to follow-up)
  evolution of comorbidities: evolution of medical treatment
number of oral medications | after surgery (up to 25 years or loss to follow-up)
  evolution of comorbidities: evolution of medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maud ROBERT, Pr, Principal Investigator — Department of Digestive Surgery, University Hospital of Edouard Herriot, Hospices Civils de Lyon
Locations (1):
- Department of Digestive Surgery, University Hospital of Edouard Herriot, Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Derived] Iceta S, Tardieu S, Nazare JA, Dougkas A, Robert M, Disse E. An artificial intelligence-derived tool proposal to ease disordered eating screening in people with obesity. Eat Weight Disord. 2021 Oct;26(7):2381-2385. doi: 10.1007/s40519-020-01076-2. Epub 2021 Jan 2. PMID 33387276